CLINICAL TRIAL: NCT03096834
Title: A 12-week Double-blind, Randomized, Multicenter Study Comparing the Efficacy and Safety of Once Monthly Subcutaneous 140 mg AMG 334 Against Placebo in Adult Episodic Migraine Patients Who Have Failed 2-4 Prophylactic Treatments (LIBERTY)
Brief Title: A Study Evaluating the Effectiveness of AMG 334 Injection in Preventing Migraines in Adults Having Failed Other Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAMG334A2301; 2016-002211-18 (EudraCT Number)
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Episodic Migraine
Keywords: Migraine; attack; headache; episodic; aura; AMG 334; CGRP receptor agonist; erenumab; adult
MeSH Terms: conditions — Migraine Disorders; Headache; Recurrence; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo DB (Placebo Comparator): Matching placebo subcutaneous injections administered every 4 weeks during Double-Blind Epoch
  Interventions: Biological: Placebo Pre-Filled Syringe (PFS)
- AMG334 140 mg DB (Experimental): AMG334 70 mg subcutaneous injections (2) administered every 4 weeks during Double-Blind Epoch
  Interventions: Biological: AMG334 (70 mg) Pre-Filled Syringe (PFS)
- AMG334 140 mg DB cont on AMG334 140 mg (Experimental): AMG334 70 mg subcutaneous injections (2) during DB continued on AMG334 140 mg in Open-Label Epoch
  Interventions: Biological: AMG334 (70 mg) Pre-Filled Syringe (PFS)
- Placebo in DB to AMG334 140 mg (Experimental): Placebo in Double-Blind Epoch (DB) switched to AMG334 140 mg in Open-Label Epoch
  Interventions: Biological: AMG334 (70 mg) Pre-Filled Syringe (PFS)

INTERVENTIONS:
Biological: AMG334 (70 mg) Pre-Filled Syringe (PFS) — Two injections of AMG 334 70 mg (equaling 140 mg total dose) will be administered via subcutaneous injection
  Arms: AMG334 140 mg DB; AMG334 140 mg DB cont on AMG334 140 mg; Placebo in DB to AMG334 140 mg
Biological: Placebo Pre-Filled Syringe (PFS) — Subcutaneous injection of matching placebo
  Arms: Placebo DB

SUMMARY:
The purpose of this study is to determine if AMG 334 is effective in treating migraines in patients who have failed other preventive migraine treatments.

DETAILED DESCRIPTION:
This study was a double blind, placebo-controlled, randomized trial in adult patients with episodic migraine. There was a screening period of 2 weeks to assess initial eligibility, and a 4-week baseline period. After randomization, participants entered the double-blind treatment epoch (DBTE) and had clinic visits for 12 weeks. All participants who completed the DBTE were eligible to enter the Open-Label Treatment Epoch (OLTE) for up to 156 weeks. All participants had a 12 week Follow-Up Epoch and a a Follow-Up visit 16 weeks after the last dose of AMG334 unless the participant continued on commercially available AMG334. Participants who had demonstrated clinical benefit were eligible to enter a Post Trial Access (PTA-Open Label Treatment Epoch) of flexible duration for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of migraine in the 12 months prior to screen
* 4-14 days per month of migraine symptoms
* >=80% diary compliance during the Baseline period
* Failure of previous migraine prophylactic treatments

Exclusion Criteria:

* >50 years old at migraine onset
* Pregnant or nursing
* History of cluster or hemiplegic headache
* Evidence of seizure or psychiatric disorder
* Score of over 19 on Beck Depression Inventory-2
* Active chronic pain syndrome
* Cardiac or hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (57):
- Novartis Investigative Site, Heidelberg, Australia
- Austria (2):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
- Czechia (3):
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, Czech Republic
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Glostrup Municipality, Denmark
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Turku
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Wiesbaden
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Glyfada
  - Novartis Investigative Site, Marousi
- Italy (6):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Palermo
- Netherlands (3):
  - Novartis Investigative Site, Sittard-Geleen, BG
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Nijmegen
- Norway (2):
  - Novartis Investigative Site, Hamar
  - Novartis Investigative Site, Sandvika
- Spain (6):
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Zaragoza
- Sweden (4):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Vällingby
- Switzerland (3):
  - Novartis Investigative Site, Bad Zurzach
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zollikon
- United Kingdom (3):
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Reuter U, Goadsby PJ, Ferrari MD, Da Silva Lima GP, Mondal S, Kalim J, Hasan F, Wen S, Arkuszewski M, Pandhi S, Stites T, Lanteri-Minet M. Efficacy and Safety of Erenumab in Participants With Episodic Migraine in Whom 2-4 Prior Preventive Treatments Had Failed: LIBERTY 3-Year Study. Neurology. 2024 May;102(10):e209349. doi: 10.1212/WNL.0000000000209349. Epub 2024 Apr 26. PMID 38669638
- [Derived] Lampl C, Kraus V, Lehner K, Loop B, Chehrenama M, Maczynska Z, Ritter S, Klatt J, Snellman J. Safety and tolerability of erenumab in individuals with episodic or chronic migraine across age groups: a pooled analysis of placebo-controlled trials. J Headache Pain. 2022 Aug 18;23(1):104. doi: 10.1186/s10194-022-01470-4. PMID 35978286
- [Derived] Ferrari MD, Reuter U, Goadsby PJ, Paiva da Silva Lima G, Mondal S, Wen S, Tenenbaum N, Pandhi S, Lanteri-Minet M, Stites T. Two-year efficacy and safety of erenumab in participants with episodic migraine and 2-4 prior preventive treatment failures: results from the LIBERTY study. J Neurol Neurosurg Psychiatry. 2022 Mar;93(3):254-262. doi: 10.1136/jnnp-2021-327480. Epub 2021 Nov 29. PMID 34845002
- [Derived] Goadsby PJ, Reuter U, Lanteri-Minet M, Paiva da Silva Lima G, Hours-Zesiger P, Fernandes C, Wen S, Tenenbaum N, Kataria A, Ferrari MD, Klatt J. Long-term Efficacy and Safety of Erenumab: Results From 64 Weeks of the LIBERTY Study. Neurology. 2021 May 31;96(22):e2724-e2735. doi: 10.1212/WNL.0000000000012029. PMID 33910942
- [Derived] Lanteri-Minet M, Goadsby PJ, Reuter U, Wen S, Hours-Zesiger P, Ferrari MD, Klatt J. Effect of erenumab on functional outcomes in patients with episodic migraine in whom 2-4 preventives were not useful: results from the LIBERTY study. J Neurol Neurosurg Psychiatry. 2021 May;92(5):466-472. doi: 10.1136/jnnp-2020-324396. Epub 2021 Jan 5. PMID 33402419
- [Derived] Reuter U, Goadsby PJ, Lanteri-Minet M, Wen S, Hours-Zesiger P, Ferrari MD, Klatt J. Efficacy and tolerability of erenumab in patients with episodic migraine in whom two-to-four previous preventive treatments were unsuccessful: a randomised, double-blind, placebo-controlled, phase 3b study. Lancet. 2018 Nov 24;392(10161):2280-2287. doi: 10.1016/S0140-6736(18)32534-0. Epub 2018 Oct 22. PMID 30360965

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 333 participants were screened for the trial
Groups:
- AMG334 140 mg DB: AMG334 140 mg subcutaneous injections administered every 4 weeks during Double-Blind Epoch
- AMG334 140 mg DB Cont on AMG334 140 mg: AMG334 140 mg subcutaneous injections during DB continued on AMG334 140 mg in Open-Label Epoch
- Placebo DB to AMG334 140 mg: Placebo in Double-Blind Epoch (DB) switched to AMG334 140 mg in Open-Label Epoch
Period: Double-Blind Treatment Epoch
Arm/Group | AMG334 140 mg DB | Placebo DB | AMG334 140 mg DB Cont on AMG334 140 mg | Placebo DB to AMG334 140 mg
Started | 121 | 125 | 0 | 0
Completed | 118 | 122 | 0 | 0
Not Completed | 3 | 3 | 0 | 0
Not completed — Protocol deviation | 2 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Subject/guardian decision | 1 | 1 | 0 | 0
Period: Open-Label Treatment Epoch
Arm/Group | AMG334 140 mg DB | Placebo DB | AMG334 140 mg DB Cont on AMG334 140 mg | Placebo DB to AMG334 140 mg
Started | 0 | 0 | 118 | 122
Completed | 0 | 0 | 86 | 83
Not Completed | 0 | 0 | 32 | 39
Not completed — Lack of Efficacy | 0 | 0 | 15 | 15
Not completed — Adverse Event | 0 | 0 | 5 | 6
Not completed — New therapy for study indication | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Subject/guardian decision | 0 | 0 | 9 | 17
Period: Safety Follow-Up Epoch
Arm/Group | AMG334 140 mg DB | Placebo DB | AMG334 140 mg DB Cont on AMG334 140 mg | Placebo DB to AMG334 140 mg
Started (After completing the Double-Blind and/or Open -Label Epoch, a Follow-Up Visit (16 weeks after the last dose of AMG334) was required as part of routine safety monitoring unless participants continued onto commercial AMG334 (contingent upon marketing authorization and commercial availability in the participating country).) | 0 | 0 | 66 | 61
Completed | 0 | 0 | 65 | 59
Not Completed | 0 | 0 | 1 | 2
Not completed — New therapy for study indication | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Period: Post-Trial Access Epoch
Arm/Group | AMG334 140 mg DB | Placebo DB | AMG334 140 mg DB Cont on AMG334 140 mg | Placebo DB to AMG334 140 mg
Started (Only participants who had demonstrated continued clinical benefit and who did not have access to commercially available drug were eligible to enter to Post-Trial Access Epoch.) | 0 | 0 | 21 | 15
Completed | 0 | 0 | 21 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG334 140 mg DB | Placebo DB | Total
Number analyzed (Participants) | 121 | 125 | 246
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 121 | 125 | 246
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 103 | 200
  Male | 24 | 22 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 112 | 115 | 227
  Asian | 0 | 1 | 1
  Unknown | 0 | 1 | 1
  Other | 9 | 8 | 17
Monthly Migraine Days at Baseline [Mean (Standard Deviation); unit: Migraine days/month] — A migraine day was defined as any calendar day in which the subject experienced a qualified migraine headache defined as: with/without aura, lasting ≥ 30 minutes with at least 1 criteria: 1. ≥ 2 of following pain features: unilateral, throbbing, moderate to severe or exacerbated with exercise/physical activity, 2. ≥ 1 of the following symptoms: nausea and/or vomiting, photophobia and phonophobia. If a migraine-specific medication (ie, triptan or ergotamine) was taken during aura, or a headache, it was counted as a migraine day regardless of duration and pain features/associated symptoms.
  Migraine days/month | 9.2 (2.56) | 9.3 (2.72) | 9.3 (2.63)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline of Monthly Migraine Days (MMD) in the Last Month (Last 4 Weeks of Treatment)
Description: A migraine day was defined as any calendar day in which the subject experienced a qualified migraine headache defined as: with/without aura, lasting ≥ 30 minutes with at least 1 criteria: 1. ≥ 2 of following pain features: unilateral, throbbing, moderate to severe or exacerbated with exercise/physical activity, 2. ≥ 1 of the following symptoms: nausea and/or vomiting, photophobia and phonophobia. If a migraine-specific medication (ie, triptan or ergotamine) was taken during aura, or a headache, it was counted as a migraine day regardless of duration and pain features/associated symptoms.
Time Frame: Baseline, Month 3 (last 4 weeks of treatment)
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | AMG334 140 mg DB | Placebo DB
Number analyzed (Participants) | 119 | 124
Percentage of participants | 30.3 | 13.7
Statistical Analysis 1: Comparison: AMG334 140 mg DB vs Placebo DB; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Adjusted for stratification factor (4-7 vs. 8-14) migraine days at Baseline after missing data are imputed as non-response (NRI); Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.43 to 5.19]

2. Secondary Outcome: Change From Baseline in Monthly Migraine Days (MMD) in the Last Month (Last 4 Weeks of Treatment)
Description: as for outcome 1
Time Frame: Baseline, Month 3 (last 4 weeks of treatment)
Population: Number of participants with both baseline and valid post baseline value from the Full Analysis Set
Measure: Mean (Standard Error); unit: Monthly migraine days
Arm/Group | AMG334 140 mg DB | Placebo DB
Number analyzed (Participants) | 118 | 120
Monthly migraine days | -1.75 (0.43) | -0.16 (0.41)
Statistical Analysis 1: Comparison: AMG334 140 mg DB vs Placebo DB; Month 3; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-2.67 to -0.51], Standard Error of Mean 0.55

3. Secondary Outcome: Change From Baseline in Physical Impairment and Everyday Activities as Measured by the Migraine Physical Function Impact Diary (MPFID) at Month 3
Description: MPFID has 2 domains: Everyday Activities, which consisted of 7 items and Physical Impairment with 5 items using a 5-point scale. Scores were summed across each domain and were then transformed and used for analyses. Transforming MPFID domain scores ranged from 0-100, where higher scores were indicative of greater migraine impact (ie, higher burden)
Time Frame: Baseline, Month 3 (last 4 weeks of treatment)
Population: Number of participants with both baseline and valid post baseline value from the Full Analysis Set
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | AMG334 140 mg DB | Placebo DB
Number analyzed (Participants) | 118 | 120
scores on a scale
  Physical impairment domain | -1.85 (0.84) | 1.61 (0.80)
  Everyday activities domain | -3.36 (0.83) | 0.55 (0.81)
Statistical Analysis 1: Comparison: AMG334 140 mg DB vs Placebo DB; Physical impairment domain; Test type: Superiority; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -3.46, 95% CI 2-sided [-5.70 to -1.23], Standard Error of Mean 1.13
Statistical Analysis 2: Comparison: AMG334 140 mg DB vs Placebo DB; Everyday activities domain; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.91, 95% CI 2-sided [-6.12 to -1.70], Standard Error of Mean 1.12

4. Secondary Outcome: Change in the Number of Monthly Acute Migraine-specific Medication Treatment Days at Month 3
Description: Number of days on which acute migraine-specific medications were used were recorded in eDiary between each monthly IP dose. Migraine-Specific medications included two categories of medications: triptan-based migraine medications and ergotamine-based migraine medications. Monthly migraine-specific medication use at baseline was the number of migraine-specific medication treatment days in the baseline period.
Time Frame: Baseline, Month 3 (last 4 weeks of treatment)
Population: Number of participants with both baseline and valid post baseline value from the Full Analysis Set
Measure: Mean (Standard Error); unit: Migraine treatment specific days/month
Arm/Group | AMG334 140 mg DB | Placebo DB
Number analyzed (Participants) | 118 | 120
Migraine treatment specific days/month | -1.25 (0.24) | 0.46 (0.28)
Statistical Analysis 1: Comparison: AMG334 140 mg DB vs Placebo DB; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.43 to -0.99], Standard Error of Mean 0.36

5. Secondary Outcome: Percentage of Participants With a 75% Reduction From Baseline of Monthly Migraine Days (MMD) in the Last Month (Last 4 Weeks of Treatment)
Description: as for outcome 1
Time Frame: Baseline, Month 3 (last 4 weeks of treatment)
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | AMG334 140 mg DB | Placebo DB
Number analyzed (Participants) | 119 | 124
Percentage of participants | 11.8 | 4.0
Statistical Analysis 1: Comparison: AMG334 140 mg DB vs Placebo DB; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel; Adjusted for stratification factor (4-7 vs. 8-14) migraine days at Baseline after missing data are imputed as non-response; Odds Ratio (OR) = 3.16, 95% CI 2-sided [1.11 to 9.01]

6. Secondary Outcome: Percentage of Participants With a 100% Reduction From Baseline of Monthly Migraine Days (MMD) in the Last Month (Last 4 Weeks of Treatment)
Description: as for outcome 1
Time Frame: Baseline, Month 3 (last 4 weeks of treatment)
Population: Full analysis set
Measure: Number; unit: Percentage of participants
Arm/Group | AMG334 140 mg DB | Placebo DB
Number analyzed (Participants) | 119 | 124
Percentage of participants | 5.9 | 0

7. Secondary Outcome: Number of Participants Who Developed Anti-AMG334 Antibodies
Description: Blood samples for immunogenicity testing were collected for the measurement of anti-AMG334 binding antibodies.
Time Frame: Baseline up to approximately 180 weeks
Measure: Number; unit: participants
Groups:
- AMG334 140 mg - All Patients: All participants who received AMG334 during trial including participants who switched from placebo
Arm/Group | AMG334 140 mg - All Patients
Number analyzed (Participants) | 238
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the first dose of study treatment through the completion of the up to 196-week trial for a maximum treatment exposure of 199 weeks (includes 4 week follow-up).
Description: Safety dataset included only those patients, who received at least one dose of study drug. Among 246 patients randomized, two patients in AMG334 and one in Placebo groups were not dosed and were not included.
Arm/Group | AMG334 140 mg DB | Placebo DB | AMG334 140 mg DB Cont on AMG334 140 mg | Placebo DB to AMG334 140 mg
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/124 | 0/118 | 0/122
Serious Adverse Events (participants affected / at risk) | 2/119 | 1/124 | 16/118 | 18/122
Other Adverse Events (participants affected / at risk) | 44/119 | 43/124 | 94/118 | 101/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG334 140 mg DB (N=119) | Placebo DB (N=124) | AMG334 140 mg DB Cont on AMG334 140 mg (N=118) | Placebo DB to AMG334 140 mg (N=122)
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | 0
Inflammation of lacrimal passage (Eye disorders) | 0 | 0 | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex hepatitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Aura (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Medication overuse headache (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 2 | 2
Status migrainosus (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG334 140 mg DB (N=119) | Placebo DB (N=124) | AMG334 140 mg DB Cont on AMG334 140 mg (N=118) | Placebo DB to AMG334 140 mg (N=122)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 8 | 6
Constipation (Gastrointestinal disorders) | 2 | 2 | 11 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 8 | 7
Nausea (Gastrointestinal disorders) | 3 | 2 | 6 | 9
Fatigue (General disorders) | 3 | 2 | 9 | 8
Influenza like illness (General disorders) | 0 | 0 | 11 | 6
Injection site haematoma (General disorders) | 1 | 2 | 2 | 7
Injection site pain (General disorders) | 7 | 7 | 8 | 8
Pyrexia (General disorders) | 1 | 0 | 8 | 7
Bronchitis (Infections and infestations) | 2 | 1 | 8 | 9
Cystitis (Infections and infestations) | 1 | 2 | 7 | 8
Gastroenteritis (Infections and infestations) | 1 | 0 | 13 | 10
Influenza (Infections and infestations) | 0 | 0 | 15 | 26
Nasopharyngitis (Infections and infestations) | 6 | 12 | 45 | 68
Rhinitis (Infections and infestations) | 0 | 0 | 6 | 5
Sinusitis (Infections and infestations) | 1 | 1 | 10 | 13
Tonsillitis (Infections and infestations) | 1 | 1 | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 9 | 7
Urinary tract infection (Infections and infestations) | 0 | 1 | 8 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 9 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 15 | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 9 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5 | 7
Dizziness (Nervous system disorders) | 3 | 2 | 5 | 7
Headache (Nervous system disorders) | 0 | 0 | 5 | 7
Migraine (Nervous system disorders) | 0 | 2 | 10 | 10
Insomnia (Psychiatric disorders) | 2 | 1 | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 10 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 13 | 6
Hypertension (Vascular disorders) | 1 | 1 | 14 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03096834/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03096834/SAP_001.pdf